CLINICAL TRIAL: NCT05418647
Title: Effect of Low Versus High Dialysate Sodium Concentration During Hemodialysis on Dialysis Recovery Time: A Prospective Randomized Clinical Trial
Brief Title: Effect of Low Versus High Dialysate Sodium Concentration During Hemodialysis on Dialysis Recovery Time
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mohamed Mamdouh Mahmoud Mohamed Elsayed , MD, Assistant professor & lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dialysate Na and DRT
Record Dates: First submitted 2022-06-10; First posted 2022-06-14 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Dialysis; Complications
Keywords: hemodialysis, recovery time, dialysate Na

STUDY DESIGN:
Intervention Model Description: This research is a single-blinded randomized clinical trial in which 40 haemodialysis patients will be randomly assigned to one of the study groups using block randomization with a ratio of 1:1.
Who Masked: Participant
Masking Description: a single blinded study as participants will be unaware about the dialysate Na each patient receives
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dialysate Na (Experimental): They will receive high dialysate sodium (Na = 141 mmol/L) for 8 weeks.
  Interventions: Other: high dialysate Na
- low dialysate Na (Experimental): They will receive low dialysate sodium (Na = 136 mmol/L) for 8 weeks.
  Interventions: Other: low dialysate Na

INTERVENTIONS:
Other: high dialysate Na — high dialysate sodium (Na = 141 mmol/L) for 8 weeks
  Arms: high dialysate Na
Other: low dialysate Na — low dialysate sodium (Na = 136 mmol/L) for 8 weeks
  Arms: low dialysate Na

SUMMARY:
This research aims to assess the effect of low versus high dialysate sodium concentration during hemodialysis on dialysis recovery time

DETAILED DESCRIPTION:
Chronic kidney disease (CKD) is a general term for heterogeneous disorders affecting the structure and function of the kidney. The variation in disease expression is partly related to the cause, pathology, severity and the rate of progression. Fatigue is a well-known and frequent symptom in HD patients with a reported association with the decrease in health-related quality of life commonly found in this population. The prevalence of fatigue ranges from 60% to as high as 97% in patients on long-term renal replacement therapy. Despite this fact, health care providers are still unaware of both its presence and severity. Several methods have been proposed as a way to assess post-HD fatigue with the "time to recover (minutes) from HD" being one of them. Lindsay et al.assisted patients' responses to the single open-ended question, "How long does it take you to recover from a dialysis session?". Although post-HD fatigue commonly exists in dialysis patients, it is usually underestimated by physicians. For this reason, appropriate and early identification of symptoms and associated factors might improve the patient's quality of life. Rayner et al. found that dialysate Na was inversely associated with DRT where lowering the Na concentration in the dialysate (to 140 mEq/L) was linked to a longer DRT.

ELIGIBILITY:
Inclusion Criteria:

* Patients with end-stage renal disease who have been prescribed long term hemodialysis and undergo four-hour HD treatments three times a week for more than 90 days.
* Patient must be at least 18 years old. They must be able to read and write, as well as be in complete mental health.

Exclusion Criteria:

* Inability to complete the surveys due to reading or hearing difficulties, actual instability of clinical condition that necessitate hospitalization, dementia, active malignancy or liver failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in dialysis recovery time | baseline, weeks 4 and 8
  By assessing the patients' responses to the single open-ended question, "How long does it take you to recover from a dialysis session?"

SECONDARY OUTCOMES:
Change in plasma sodium concentration | baseline, weeks 4 and 8
  measuring plasma sodium concentration
Change in the inter-dialytic weight gain | 8 weeks
  measuring the inter-dialytic weight gain
Change in blood pressure (systolic, diastolic, mean) | 8 weeks
  measuring in blood pressure (systolic, diastolic, mean)
Occurrence of intradialytic hypotension | 8 weeks
  incidence of intradialytic hypotension
Occurrence of muscle cramps | 8 weeks
  incidence of muscle cramps
Occurrence of headache | 8 weeks
  incidence of headache

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Mamdouh Elsayed, MD, Principal Investigator — lecturer; osama M Refai, MBBCh, Study Chair — resident of Nephrology & Internal Medicine, Alexandria University Hospitals
Locations (2):
- Egypt (2):
  - Faculty of Medicine, Aexandria University, Alexandria
  - Faculty of Medicine, Alexandria University, Alexandria

REFERENCES:
- [Background] Levey AS, Stevens LA, Coresh J. Conceptual model of CKD: applications and implications. Am J Kidney Dis. 2009 Mar;53(3 Suppl 3):S4-16. doi: 10.1053/j.ajkd.2008.07.048. PMID 19231760
- [Background] Murtagh FE, Addington-Hall J, Higginson IJ. The prevalence of symptoms in end-stage renal disease: a systematic review. Adv Chronic Kidney Dis. 2007 Jan;14(1):82-99. doi: 10.1053/j.ackd.2006.10.001. PMID 17200048
- [Background] Weisbord SD, Fried LF, Arnold RM, Fine MJ, Levenson DJ, Peterson RA, Switzer GE. Prevalence, severity, and importance of physical and emotional symptoms in chronic hemodialysis patients. J Am Soc Nephrol. 2005 Aug;16(8):2487-94. doi: 10.1681/ASN.2005020157. Epub 2005 Jun 23. PMID 15975996
- [Background] Weisbord SD, Fried LF, Mor MK, Resnick AL, Unruh ML, Palevsky PM, Levenson DJ, Cooksey SH, Fine MJ, Kimmel PL, Arnold RM. Renal provider recognition of symptoms in patients on maintenance hemodialysis. Clin J Am Soc Nephrol. 2007 Sep;2(5):960-7. doi: 10.2215/CJN.00990207. Epub 2007 Aug 8. PMID 17702730
- [Background] Lindsay RM, Heidenheim PA, Nesrallah G, Garg AX, Suri R; Daily Hemodialysis Study Group London Health Sciences Centre. Minutes to recovery after a hemodialysis session: a simple health-related quality of life question that is reliable, valid, and sensitive to change. Clin J Am Soc Nephrol. 2006 Sep;1(5):952-9. doi: 10.2215/CJN.00040106. Epub 2006 Jul 6. PMID 17699312
- [Background] Rayner HC, Zepel L, Fuller DS, Morgenstern H, Karaboyas A, Culleton BF, Mapes DL, Lopes AA, Gillespie BW, Hasegawa T, Saran R, Tentori F, Hecking M, Pisoni RL, Robinson BM. Recovery time, quality of life, and mortality in hemodialysis patients: the Dialysis Outcomes and Practice Patterns Study (DOPPS). Am J Kidney Dis. 2014 Jul;64(1):86-94. doi: 10.1053/j.ajkd.2014.01.014. Epub 2014 Feb 14. PMID 24529994